CLINICAL TRIAL: NCT05657873
Title: A Phase II Trial of Hepatic Ablation of Metastases to Modulate and Enhance Immunotherapy Response (HAMMER) in NSCLC
Brief Title: A Study of Targeted Radiation Therapy in People With Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-386
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Non-small Cell Carcinoma; NSCLC; NSCLC Stage IV
Keywords: non small cell lung cancer; Non Small Cell Lung Cancer Metastatic; Non-small Cell Carcinoma; liver stereotactic ablative radiotherapy; L-SABR; NSCLC; NSCLC Stage IV; Memorial Sloan Kettering Cancer Center; 22-368
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- L-SABR Arm (Experimental): Participants randomized to the experimental arm will continue with standard of care treatment but will also undergo radiation simulation for L-SABR/Liver Stereotactic Ablative Radiation Therapy.
  Interventions: Radiation: L-SABR; Biological: Anti-PD-(L)1 based immunotherapy; Drug: Platinum based chemotherapy
- Control Arm (Active Comparator): Participants randomized to the control arm will be treated according to the standard of care.
  Interventions: Biological: Anti-PD-(L)1 based immunotherapy; Drug: Platinum based chemotherapy

INTERVENTIONS:
Radiation: L-SABR — L-SABR will be delivered in a week during which the patient receives no chemotherapy. L-SABR can be on the same week or even day as anti-PD-(L)1 therapy.
  Other Names: Liver Stereotactic Ablative Radiation Therapy
  Arms: L-SABR Arm
Biological: Anti-PD-(L)1 based immunotherapy — Standard of care treatment (anti-PD-(L)1 based immunotherapy +/- platinum based chemotherapy
  Other Names: Standard of Care
Drug: Platinum based chemotherapy — Standard of care treatment (anti-PD-(L)1 based immunotherapy +/- platinum based chemotherapy
  Other Names: Standard of Care

SUMMARY:
The purpose of this study is to see whether adding liver stereotactic ablative radiotherapy/L-SABR to standard drug therapy is better than standard drug therapy alone for people with metastatic non-small cell lung cancer/NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Be greater than 18 years of age on day of signing informed consent.
* Have a histologically confirmed diagnosis of stage IV NSCLC (includes patients who have progressed on durvalumab for Stage III NSCLC) without known mutations in (EGFR) or BRAF or rearrangements in ALK (anaplastic lymphoma kinase) or ROS-1.
* Newly diagnosed metastatic non-small cell lung cancer (NSCLC), including both de novo and secondary metastatic disease, with one or more liver metastases
* Plan to initiate standard of care anti-PD-(L)1 based immunotherapy +/- platinum based chemotherapy for at least 3 cycles

  o Regimens combining anti-CTLA-4 immunotherapy with anti-PD-1 (e.g., ipilimumab plus nivolumab) or anti-PD-L1 (e.g., tremelimumab plus durvalumab) immunotherapy are allowed.
* Have a performance status of 0-2 on the ECOG Performance Scale.
* Liver function tests:

  * Total Bilirubin ≤ 1.5 x ULN
  * AST/ ALT ≤ 5 x ULN
* Eligible for L- SABR to all liver metastases.
* Patients with known HIV are eligible provided they are under treatment with effective anti-retroviral therapy with CD4 >200 cells/microliter ≤ 28 days prior to registration

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.
* Patients with prior external beam radiation therapy to the liver.
* Patients with known active Hepatitis B or Hepatitis C.
* Patients with immunosuppression including pharmacological immunosuppression with chronic steroids or immune modulators like cyclosporin or methotrexate and patients with active autoimmune disease.
* Patients who are pregnant or breastfeeding
* Men or women not using effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival | up to 4 years
  Primary outcomes is to determine if L-SABR, when added to first line standard of care anti-PD-(L)1 based immunotherapy +/- chemotherapy, can improve median progression-free survival (PFS) in patients with metastatic NSCLC involving the liver.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Romesser, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - BAPTIST ALLIANCE - MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] McMillan MT, Reyngold M, Crane CH, O'Brien DAR, Williams VM, Zinovoy M, Cuaron JJ, Gonen M, Kaiser A, Sopka DM, Gomez DR, Schoenfeld AJ, Bott M, Romesser PB. A phase II trial of hepatic ablation of metastases to modulate and enhance immunotherapy response in non-small cell lung cancer (HAMMER-NSCLC). BMC Cancer. 2025 Sep 2;25(1):1408. doi: 10.1186/s12885-025-14779-5. PMID 40898159
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org